CLINICAL TRIAL: NCT00000711
Title: Granulocyte-Macrophage Colony-Stimulating Factor and Zidovudine: A Phase I Study of Concurrent Administration in Patients With AIDS and Severe ARC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 065; 11039 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Cytopenias
Keywords: Neutropenia; Drug Evaluation; Drug Therapy, Combination; Granulocyte-Macrophage Colony-Stimulating Factor; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Cytopenia; Neutropenia; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine; sargramostim

INTERVENTIONS:
Drug: Zidovudine
Drug: Sargramostim

SUMMARY:
To administer colony-stimulating factor (GM-CSF) for 4 weeks to AIDS and advanced AIDS related complex (ARC) patients who have been receiving zidovudine (AZT) therapy, in order to obtain data on short-term effectiveness, safety, toxicity, pharmacokinetics, and tolerance of combined treatment with the two drugs.

Persons infected with HIV virus may undergo a long latency or persistent virus blood levels which may be present before any symptomatic illness. These individuals could, therefore, benefit from therapy with an effective antiretroviral agent. AZT, which is a powerful inhibitor of human retrovirus, has been approved for management of patients with symptomatic HIV infection. GM-CSF not only stimulates the bone marrow, it enhances the function of mature blood cells and has been found to enhance the ability of AZT to suppress HIV replication in vitro (test tube). Combination therapy with GM-CSF and AZT may lower complications as well as the morbidity and mortality associated with HIV infection.

DETAILED DESCRIPTION:
Persons infected with HIV virus may undergo a long latency or persistent virus blood levels which may be present before any symptomatic illness. These individuals could, therefore, benefit from therapy with an effective antiretroviral agent. AZT, which is a powerful inhibitor of human retrovirus, has been approved for management of patients with symptomatic HIV infection. GM-CSF not only stimulates the bone marrow, it enhances the function of mature blood cells and has been found to enhance the ability of AZT to suppress HIV replication in vitro (test tube). Combination therapy with GM-CSF and AZT may lower complications as well as the morbidity and mortality associated with HIV infection.

Colony stimulating factor (GM-CSF) is administered subcutaneously, once a day or every other day, for 4 weeks to AIDS and advanced ARC patients who have been receiving and will continue to receive a constant dose of AZT. Treatment is on an outpatient basis.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Modest doses of acetaminophen, aspirin, or non-prescription doses of ibuprofen may be used with caution for fever control and mild analgesia. Prolonged use more than 72 hours is not advised without dose supervision.

All patients should have a documented history of positive HIV antibody by ELISA test. Patients should qualify for zidovudine (AZT) treatment for the following reasons:

* Patients with a prior episode of cytologically confirmed Pneumocystis carinii pneumonia (PCP).
* Patients with a prior episode of any AIDS-defining opportunistic infection and less than 200 T4 cells.
* Patients with advanced ARC as defined by mucocutaneous candidiasis and/or unexplained weight loss and less than 200 T4 cells and fever more than 100 degrees F of more than 3 weeks duration; clinical diagnosis of hairy leukoplakia; herpes zoster infection within 3 months of entry; or unexplained diarrhea.
* All patients must have received at least 8 weeks of AZT prior to enrollment and must not have required a dose adjustment for the previous 4 weeks.
* Patients must be willing to sign an informed consent statement.

Required:

* Zidovudine (AZT) for at least 8 weeks.

Exclusion Criteria

Co-existing Condition:

The following patients will be excluded:

* Patients receiving zidovudine (AZT) while enrolled in another protocol.
* Patients with other life-threatening and uncontrolled opportunistic infection.
* Patients with evidence of lymphoma or neoplasm other than indolent Kaposi's sarcoma.
* Dementia that would prevent giving appropriate informed consent.

Concurrent Medication:

Excluded:

* Acetaminophen or products containing acetaminophen.
* Drugs that are nephrotoxic, are cytotoxic, or decrease blood cell number or function may increase the risk of toxicity.

Probenecid may inhibit excretion of zidovudine (AZT). Some experimental nucleoside analogs should be avoided.

The following patients will be excluded:

* Patients receiving zidovudine (AZT) while enrolled in another protocol.
* Patients with other life-threatening and uncontrolled opportunistic infection.
* Patients with evidence of lymphoma or neoplasm other than indolent Kaposi's sarcoma.
* Dementia that would prevent giving appropriate informed consent.

Prior Medication:

Excluded within 8 weeks of study entry:

* Prior systemic therapy with an antimetabolite, cytotoxic drug, interferon, immunomodulator, corticosteroid, or nucleoside analog other than zidovudine.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Study Completion 1990-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hewitt RG, Study Chair
Locations (1):
- SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York, United States

REFERENCES:
- [Background] Portmore A, Morse G, Hewitt R, Reichman R. Comparative oral disposition of zidovudine in neutropenic AIDS patients and asymptomatic hemophiliacs. Int Conf AIDS. 1990 Jun 20-23;6(3):196 (abstract no SB442)
- [Background] Hewitt RG, Morse GD, Lawrence WD, Maliszewski ML, Santora J, Bartos L, Bonnem E, Poiesz B. Pharmacokinetics and pharmacodynamics of granulocyte-macrophage colony-stimulating factor and zidovudine in patients with AIDS and severe AIDS-related complex. Antimicrob Agents Chemother. 1993 Mar;37(3):512-22. doi: 10.1128/AAC.37.3.512. PMID 8460920
- [Derived] Wang GJ, Zhao J, Tomasi D, Kojori ES, Wang R, Wiers CE, Caparelli EC, Volkow ND. Effect of combined naltrexone and bupropion therapy on the brain's functional connectivity. Int J Obes (Lond). 2018 Nov;42(11):1890-1899. doi: 10.1038/s41366-018-0040-2. Epub 2018 Feb 23. PMID 29535451